CLINICAL TRIAL: NCT03769142
Title: Cerebral Perfusion Changes During General Anesthesia Induction: Relation Between Transcranial Doppler, Bispectral Index and Cerebral Oximetry: a Prospective Observational Study
Brief Title: Cerebral Perfusion During Induction of General Anesthesia
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); Department of Anesthesiology, Hopital Foch, Suresnes, France. (Unknown); M3DISIM (Other); Ouctomes Research Consortium, Cleveland Clinic, Ohio, USA (Unknown)
Responsible Party: Sponsor
Other Study IDs: SRLF 11-356
Record Dates: First submitted 2018-10-10; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-10

CONDITIONS: Radiography; Interventional
Keywords: cerebral perfusion; hypotension; transcranial Doppler; general anesthesia; Bispectral Index; Near-infrared spectroscopy (NIRS)
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: All monitoring — All monitoring (TCD, BIS, NIRS) are collected from the healthy side, contralateral to the interventional side

SUMMARY:
Arterial hypotension during general anesthesia remains a factor of poor outcomes, increases the risk of myocardial infarction, acute kidney injury and 1-year mortality. Furthermore, arterial hypotension may also decrease cerebral perfusion contributing to worsen neurological outcome. It seems necessary to monitor cerebral perfusion during anesthesia and to define individual dynamic targets of blood pressure. The goal of this study is to evaluate cerebral perfusion change in adult patients with or without cardiovascular risk factors during a standardized propofol-remifentanil anesthesia induction. Cerebral perfusion will be evaluated and compared using the simultaneously measure of TCD, NIRS and BIS. Those measures will be also repeated during and after treatment of arterial hypotension episodes in both groups.

DETAILED DESCRIPTION:
Main objective : the blood pressure target to maintain cerebral perfusion is related to patient´s characteristics or comorbidities and it remains uncertain which threshold of blood pressure to use during general anesthesia. Thus, it seems necessary to monitor cerebral perfusion during anesthesia and to define individual dynamic targets of blood pressure. The measure of middle cerebral artery blood flow velocity by transcranial doppler (TCD) is a clinical method to assess cerebral perfusion during general anesthesia and several studies have reported the hemodynamic impact on cerebral blood flow during induction.

Cerebral perfusion can also be approached by near infrared spectroscopy (NIRS) which measures continuously cerebral oxygen saturation.

Bispectral index (BIS) which allows a simplified form of continuous electroencephalogram monitoring to assess depth of anesthesia could also report cerebral hypoperfusion quantified by the count of burst suppression ratio (SR). Potentially, those tools need to be combined to assess cerebral perfusion properly.

The goal of this study is to evaluate cerebral perfusion change in adult participants with or without cardiovascular risk factors during a standardized propofol-remifentanil anesthesia induction. Cerebral perfusion was evaluated and compared using the simultaneously measure of TCD, NIRS and BIS. Those measures will be also repeated during and after treatment of arterial hypotension episodes in both groups.

Experimental design : this is a single-center, interventional, category II prospective study (minimal risks and constraints) Population concerned :the study involves major patients who beneficiate from intraoperative hemodynamic optimization with norepinephrine (as noradrenaline tartrate) for maintaining blood pressure under general anaesthesia in interventional neuroradiology in adults.

Research Proceedings : all monitoring (TCD, BIS, NIRS) are collected from the healthy side, contralateral to the interventional side. BIS, NIRS and continuous non-invasive blood pressure are all connected to the main monitor. For all participants, data from TCD, NIRS, BIS and hemodynamic data are collected at three distinct periods the day of the procedure : (1) baseline or during pre-oxygenation at FiO2 21% (inspiratory fraction oxygen) in awake patients, (2) before Orotracheal Intubation and (3) just after mechanical ventilation.

In patients presenting a hypotensive episode at any time of the procedure, all parameters are collected before and at the peak effect of a 10µg bolus of norepinephrine Individual benefit:there is no benefit for the patient

Collective benefit: It seems necessary to monitor cerebral perfusion during anesthesia and to define individual dynamic targets of blood pressure. During general anesthesia, cerebral perfusion can be impaired and requires specific monitoring.

Risks and minimal constraints added by the research : no added risk. This clinical research work is "non-interventional" on adult patients who benefit from a neuroradiological intervention. All measures are obtained non-invasively.

Patients were assigned to one of two groups according to cardiovascular risk factors. Major risk factor was age > 50 years old and minor risk factors were history of congestive heart failure, history of cardiovascular event, current smoking, diabetes mellitus, dyslipidemia, arterial hypertension.

Patients will be classified into the high-risk group (Hi-risk) if they have at least one major criterion or two minor criteria or into the low risk group (Lo-risk) if they present with no or one minor criterion.

During their interventional neuroradiology procedure, all patients' routine monitoring will consist of electrocardiogram, pulsated oxygen saturation, end-tidal C02 (carbon dioxide), respiratory rate, tidal volume and monitoring of neuromuscular function.

For all patients whatever the comorbidities, anesthesia induction will be performed using a target-controlled infusion (Orchestra® Base Primea - Fresenius Kabi France).

According to our standard of care, intra-operative episodes of hypotension (mean arterial pressure (MAP) < 65 mmHg or < 80% baseline) were treated by Norepinephrine bolus of 10 µg.

For all patients, data from TCD, NIRS, BIS and hemodynamic data will be collected at three distinct periods: (1) Baseline or during pre-oxygenation at FiO2 21% (Inspiratory Fraction Oxygen) in awake patients, (2) Before Orotracheal Intubation and (3) just after mechanical ventilation.

In patients presenting a hypotensive episode at any time of the procedure, all parameters were collected before and at the peak effect of a 10µg bolus of norepinephrine.

Number of selected subjects : Selection of patients up to 100 analysable patients Number of Centre : 1 Research Agenda inclusion period: 24 months Duration of participation (treatment + follow-up): duration of the interventional neuroradiology procedure so maximum 1 day Total duration: 24 months Number of planned inclusions by centre and month : 5 Number of subjects required : 100

Statistics

Changes of parameters across time, during induction and/or during vasopressors boluses will be tested by using a paired Student-t test after testing the normality of distribution. Correlation between change of MAP and Vm during induction will be done using Spearman test. Complete analysis will also be performed and compared between Low-risk and High-risk patients. The analysis of vasopressor boluses will also be performed according to the time of the administration: boluses which are given immediately after induction of anesthesia (early) and boluses given after a 30 minutes period of constant intra-venous calculated concentrations of anesthesia (late). All statistical analyses were performed using R statistical software (The 'R' Foundation for Statistical Computing, Vienna, Austria). Results are expressed as means (± SD). A two-sided p value of 0.05 was considered significant.

The sample size calculation is based on the following assumptions: incidence of Hi-risk patients of 50%, as previously reported, incidence of burst suppression during induction in low risk patients of 20% difference of incidence of burst suppression between low- and high-risk patients at 30%, power at 80% and type I error at 5%. Accordingly, the calculated sample size is 100 patients for the entire population.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years, scheduled an elective interventional neuroradiology procedure requiring general anesthesia
* oral agreement obtained from each patient before anesthesia

Exclusion Criteria:

* age <18 years
* an emergency procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with scheduled an elective interventional neuroradiology procedure requiring general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Continuous measure of mean arterial pressure in mmHg (MAP) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, mean arterial pressure will be collected at three distinct periods: (1) Baseline or during pre-oxygenation at FiO2 21% in awake patients, (2) Before Orotracheal Intubation and (3) just after mechanical ventilation
Measure of cerebral blood flow (CFV in cm/s) with Transcranial Doppler | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, cerebral flow velocity will be collected at three distinct periods: (1) Baseline or during pre-oxygenation at FiO2 21% in awake patients, (2) Before Orotracheal Intubation and (3) just after mechanical ventilation.
Continuous measure of Burst Suppression (BS in %) with Bispectral Index (BIS) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, Burst Supression will be collected at three distinct periods: (1) Baseline or during pre-oxygenation at FiO2 21% in awake patients, (2) Before Orotracheal Intubation and (3) just after mechanical ventilation.
Continuous measure of cerebral oxygen saturation (SO2 in %) with Near-infrared spectroscopy (NIRS) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, cerebral oxygen saturation will be collected at three distinct periods: (1) Baseline or during pre-oxygenation at FiO2 21% in awake patients, (2) Before Orotracheal Intubation and (3) just after mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MATEO, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Manquat E, Ravaux H, Kindermans M, Joachim J, Serrano J, Touchard C, Mateo J, Mebazaa A, Gayat E, Vallee F, Cartailler J. Impact of impaired cerebral blood flow autoregulation on electroencephalogram signals in adults undergoing propofol anaesthesia: a pilot study. BJA Open. 2022 Mar 2;1:100004. doi: 10.1016/j.bjao.2022.100004. eCollection 2022 Mar. PMID 37588691